CLINICAL TRIAL: NCT02717442
Title: A Prospective, Randomized, Double-blind, Placebo-controlled, Multicenter, Phase 3 Study of OTO-104 Given as a Single Intratympanic Injection in Subjects With Unilateral Meniere's Disease
Brief Title: Study of OTO-104 in Subjects With Unilateral Meniere's Disease
Acronym: AVERTS-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Negative Efficacy Results from the recently completed Phase 3 study 104-201506
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 104-201508
Record Dates: First submitted 2016-03-10; First posted 2016-03-23 (Estimated); Results first posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-12

CONDITIONS: Meniere's Disease
Keywords: Meniere's Disease; Vertigo
MeSH Terms: conditions — Meniere Disease; Vertigo

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OTO-104 (Experimental): 12 mg dexamethasone
  Interventions: Drug: OTO-104
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OTO-104 — Single intratympanic injection of 12 mg OTO-104
  Arms: OTO-104
Drug: Placebo — Single intratympanic injection of placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of OTO-104 for the treatment of Meniere's disease.

ELIGIBILITY:
Inclusion Criteria includes, but is not limited to:

* Subject has a diagnosis of unilateral Meniere's disease by 1995 American Academy of Otolaryngology - Head and Neck Surgery (AAOHNS) criteria and reports active vertigo for the 2 months prior to the study lead-in period.
* Subject has experienced active vertigo during the lead-in period.
* Subject has documented asymmetric sensorineural hearing loss.
* Subject agrees to maintain their current treatments for Meniere's disease while on-study.

Exclusion Criteria includes, but is not limited to:

* Subject is pregnant or lactating.
* Subject has a history of immunodeficiency disease.
* Subject has a history of previous endolymphatic sac surgery.
* Subject has a history of previous use of intratympanic (IT) gentamicin in the affected ear.
* Subject has a history of tympanostomy tubes with evidence of perforation or lack of closure.
* Subject has experienced an adverse reaction to IT injection of steroids.
* Subject has used an investigational drug or device in the 3 months prior to screening.
* Subject has previously been randomized to a trial of OTO-104.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathie Bishop, PhD, Study Chair — Otonomy, Inc.
Locations (1):
- Many sites in Europe. Refer to the contact info listed below., San Diego, California, United States

REFERENCES:
- [Derived] Phillips J, Mikulec AA, Robinson JM, Skarinsky D, Anderson JJ. Efficacy of Intratympanic OTO-104 for the Treatment of Meniere's Disease: The Outcome of Three Randomized, Double-Blind, Placebo-Controlled Studies. Otol Neurotol. 2023 Jul 1;44(6):584-592. doi: 10.1097/MAO.0000000000003886. Epub 2023 Apr 22. PMID 37185596

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 176 subjects were randomized and 174 subjects received study drug. The most common reason for screen failure was insufficient number of definitive vertigo days in the 28-day lead-in period. The first subject enrolled March 21, 2016, and the last subject completed September 15, 2017. A total of 49 centers in Europe (Belgium, France, Germany, Italy, Poland, United Kingdom) enrolled subjects.
Pre-assignment Details: This study was terminated early based on results of study 104-201506, a US Phase 3 study that indicated no statistically significant difference in the primary endpoint of reduction in definitive vertigo days (DVD) for OTO-104 vs placebo nor for any of the secondary endpoints. Decision was made to terminate all ongoing studies on August 31, 2017, including this study. At the time of termination, 112/176 randomized subjects completed the study out to Week 12 (Month 3).
Period: Overall Study
Arm/Group | OTO-104 | Placebo
Started | 88 | 88
Completed | 53 | 59
Not Completed | 35 | 29
Not completed — Study Terminated by Sponsor | 31 | 29
Not completed — Subject Randomized, but Did not Receive Drug | 2 | 0
Not completed — Other - Not Specified | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- OTO-104 (Full Analysis Set -1): Subjects that were randomized to OTO-104, received study drug, had a baseline definitive vertigo measurement (i.e., at least 1 baseline daily diary entry) for the 4-week lead-in period and at least one 4-week definitive vertigo measurement post-baseline (i.e., at least 1 post baseline daily diary entry).
- Placebo (Full Analysis Set - 1): Subjects that were randomized to placebo, received study drug, had a baseline definitive vertigo measurement(i.e., at least 1 baseline daily diary entry) for the 4-week lead-in period and at least one 4-week definitive vertigo measurement post-baseline (i.e., at least1 post baseline daily diary entry).
- Total: Total of all reporting groups
Arm/Group | OTO-104 (Full Analysis Set -1) | Placebo (Full Analysis Set - 1) | Total
Number analyzed (Participants) | 86 | 88 | 174
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 75 | 147
  >=65 years | 14 | 13 | 27
Age, Continuous [Median (Full Range); unit: years] | 53.0 [19 to 81] | 53.0 [22 to 80] | 53.0 [19 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 48 | 92
  Male | 42 | 40 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 77 | 75 | 152
  Unknown or Not Reported | 9 | 12 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 82 | 82 | 164
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  Belgium | 3 | 5 | 8
  France | 4 | 5 | 9
  Germany | 13 | 15 | 28
  Italy | 12 | 6 | 18
  Poland | 28 | 34 | 62
  United Kingdom | 26 | 23 | 49
Previous IT Steroid Injection [Count of Participants; unit: Participants] | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: The Number of DVD at Week 12 (the 4-week [28 Days] Interval From Week 9 Through Week 12) - FAS-1 Population
Description: In the Full Analysis Set (FAS)-1 population, the number of DVDs at Week 12 (the 4-week [28 days] interval from Week 9 through Week 12) was compared between OTO-104 and placebo. Week 12 = 12 weeks after dosing at the Baseline visit. The Baseline visit occurred at the end of lead-in. No intervention was administered during lead-in.
Time Frame: 3 months
Population: A subject is included in the analysis if they received study drug, had a baseline definitive vertigo measurement for the 4-week lead-in period and at least one 4-week definitive vertigo measurement post-baseline, i.e., at least one post-baseline daily diary entry. The model and corresponding method of estimation adjusted for overdispersion and addressed missing 4-week intervals under the assumption of Missing at Random (MAR).
Measure: Mean (95% Confidence Interval); unit: Definitive Vertigo Day
Groups:
- Placebo (Full Analysis Set - 1): Subjects that were randomized to placebo, received study drug, had a baseline definitive vertigo measurement (i.e., at least 1 baseline daily diary entry) for the 4-week lead-in period and at least one 4-week definitive vertigo measurement post-baseline (i.e., at least 1 post baseline daily diary entry).
Arm/Group | OTO-104 (Full Analysis Set -1) | Placebo (Full Analysis Set - 1)
Number analyzed (Participants) | 86 | 88
Definitive Vertigo Day | 2.336 [1.747 to 3.125] | 3.549 [2.763 to 4.560]
Statistical Analysis 1: Comparison: OTO-104 (Full Analysis Set -1) vs Placebo (Full Analysis Set - 1); The primary efficacy endpoint was compared between OTO-104 and placebo at the 2-tailed 0.05 alpha level using a generalized Poisson linear mixed model. The model included fixed effects for randomized treatment group, sex, study week, a treatment group by study week interaction, and the count of lead-in period DVD standardized to 28 days as a covariate; Test type: Superiority; p = 0.029, Regression, Linear — Study week was based on each 4-week interval and was modeled as a categorical variable, and an offset for the log of the number of diary entries recorded for each 4-week interval post-baseline was included for each subject; Risk Ratio (RR) = 0.658, 95% CI 2-sided [0.453 to 0.957]

2. Primary Outcome: The Number of DVD at Week 12 (the 4-week [28 Days] Interval From Week 9 Through Week 12) - FAS-2 Population
Description: The number of DVDs at Week 12 (the 4-week [28 days] interval from Week 9 through Week 12) was compared between OTO-104 and placebo. Week 12 = 12 weeks after dosing at the Baseline visit. The Baseline visit occurred at the end of lead-in. No intervention was administered during lead-in.
Time Frame: 3 months
Population: The FAS - 2 includes all subjects from FAS-1 who were randomized 12 weeks prior to the study termination decision date of August 31, 2017 (i.e., subjects that had the opportunity to complete 12 weeks of daily diary entries in the study at the time of study termination).
Measure: Mean (95% Confidence Interval); unit: Definitive Vertigo Day
Groups:
- OTO-104 (Full Analysis Set -2): Subjects in the FAS-1 that were randomized to OTO-104 12 weeks prior to the study termination decision date of August 31, 2017 (i.e., subjects that had the opportunity to complete 12 weeks of daily diary entries in the study at the time of study termination)
- Placebo (Full Analysis Set - 2): Subjects in the FAS-1 that were randomized to Placebo 12 weeks prior to the study termination decision date of August 31, 2017 (i.e., subjects that had the opportunity to complete 12 weeks of daily diary entries in the study at the time of study termination)
Arm/Group | OTO-104 (Full Analysis Set -2) | Placebo (Full Analysis Set - 2)
Number analyzed (Participants) | 55 | 56
Definitive Vertigo Day | 2.044 [1.480 to 2.822] | 3.467 [2.617 to 4.594]
Statistical Analysis 1: Comparison: OTO-104 (Full Analysis Set -2) vs Placebo (Full Analysis Set - 2); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.014, Regression, Linear; Risk Ratio (RR) = 0.590, 95% CI 2-sided [0.388 to 0.896]

3. Secondary Outcome: Effect of Vertigo on Daily Activities - Number of Days Sick at Home or Bedridden at Week 12 (Month 3): FAS-1
Description: Week 12 = 12 weeks after dosing at the Baseline visit. The Baseline visit occurred at the end of lead-in. No intervention was administered during lead-in.
  Questionnaire - subjects were instructed to record the effect on their daily activities of their total vertigo experienced that day using a 5-point scoring system:
  0 = normal activity
  1. = slight limitation
  2. = moderate limitation
  3. = sick at home
  4. = bedridden
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Groups:
- Placebo (Full Analysis Set - 1): Subjects that were randomized to placebo, received study drug, had a baseline definitive vertigo measurement (i.e., at least 1baseline daily diary entry) for the 4-week lead-in period and at least one 4-week definitive vertigo measurement post-baseline (i.e., at least 1 post baseline daily diary entry).
Arm/Group | OTO-104 (Full Analysis Set -1) | Placebo (Full Analysis Set - 1)
Number analyzed (Participants) | 86 | 88
days | 1.2 (2.32) | 2.3 (4.58)

4. Secondary Outcome: Effect of Vertigo on Daily Activities - Number of Days Sick at Home or Bedridden at Week 12 (Month 3): FAS-2
Description: as for outcome 3
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: days
Groups:
- OTO-104 (Full Analysis Set- 2): The FAS - 2 includes subjects in the FAS-1 randomized to OTO-104 12 weeks prior to the study termination decision date of31AUG2017 (i.e., subjects that had the opportunity to complete 12 weeks of daily diary entries in the study at the time of study termination).
- Placebo (FAS-2): The FAS - 2 includes subjects in the FAS-1 randomized to Placebo 12 weeks prior to the study termination decision date of31AUG2017 (i.e., subjects that had the opportunity to complete 12 weeks of daily diary entries in the study at the time of study termination).
Arm/Group | OTO-104 (Full Analysis Set- 2) | Placebo (FAS-2)
Number analyzed (Participants) | 55 | 56
days | 1.2 (2.18) | 2.2 (4.68)

5. Secondary Outcome: Otoscopic Examination - Tympanic Membrane Perforation at Week 12 (Month 3)
Description: Otoscopic examinations were conducted at each visit. It was considered important to understand if the tympanic perforation that resulted from the IT injection at the Baseline visit persisted at the end of study visit (Week12 [Month 3]). Week 12 = 12 weeks after dosing at the Baseline visit. The Baseline visit occurred at the end of lead-in. No intervention was administered during lead-in.
Time Frame: 3 months
Population: Only subjects that had a Month 3 otoscopic examination are included in assessment of this emdpoint.
Measure: Count of Participants; unit: Participants
Groups:
- OTO-104 (Safety Analysis Set): All subjects who receivedOTO-104. Subjects were included in this treatment group according to the actual treatment received regardless of their randomized assignment.
- Placebo (Safety Analysis Set): All subjects who received Placebo. Subjects were included in this treatment group according to the actual treatment received regardless of their randomized assignment.
Arm/Group | OTO-104 (Safety Analysis Set) | Placebo (Safety Analysis Set)
Number analyzed (Participants) | 53 | 59
Participants | 1 | 0

6. Secondary Outcome: Audiometry - Shift in Air-Bone Gap at 500 Hz From Baseline to Week 12 (Month 3)
Description: The number of subjects with a change in air-bone gap from Baseline to Week 12 (Month 3) from no impairment (<=10 dB) to impairment (>10 dB) when measure at 500 Hz. Week 12 = 12 weeks after dosing at the Baseline visit. The Baseline visit occurred at the end of lead-in. No intervention was administered during lead-in.
Time Frame: 3 Months
Population: Subjects that had no impairment at the baseline visit (air-bone gap <=10 dB) and had an audiogram collected at the Week 12 (Month 3) visit.
Measure: Count of Participants; unit: Participants
Arm/Group | OTO-104 (Safety Analysis Set) | Placebo (Safety Analysis Set)
Number analyzed (Participants) | 48 | 52
Participants | 8 | 7

7. Secondary Outcome: Audiometry - Shift in Air-Bone Gap at 1000 Hz From Baseline to Week 12 (Month 3)
Description: The number of subjects with a change in air-bone gap from Baseline to Week 12 (Month 3) from no impairment at baseline (<= 10 dB) to impairment at Month 3 (>10 dB) when measured at 1000 Hz. Week 12 (Month 3) = 12 weeks after dosing at the Baseline visit. The Baseline visit occurred at the end of lead-in. No intervention was administered during lead-in.
Time Frame: 3 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | OTO-104 (Safety Analysis Set) | Placebo (Safety Analysis Set)
Number analyzed (Participants) | 39 | 45
Participants | 11 | 3

8. Secondary Outcome: Audiometry - Shift in Air-Bone Gap at 2000 Hz From Baseline to Week 12 (Month 3)
Description: The number of subjects with a change in air-bone gap from Baseline to Week 12 (Month 3) from no impairment at baseline (<= 10 dB) to impairment at Month 3 (>10 dB) when measured at 2000 Hz. Week 12 (Month 3) = 12 weeks after dosing at the Baseline visit. The Baseline visit occurred at the end of lead-in. No intervention was administered during lead-in.
Time Frame: 3 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | OTO-104 (Safety Analysis Set) | Placebo (Safety Analysis Set)
Number analyzed (Participants) | 42 | 51
Participants | 0 | 4

ADVERSE EVENTS:
Time Frame: Reported or observed during or after dosing with the study drug at the Baseline visit up until the Week 12 (3 Months) end of study visit. The Baseline visit occurred at the end of lead-in. No intervention was administered during lead-in, which is why adverse events were collected starting at the Baseline visit during dosing up until the final visit.
Arm/Group | OTO-104 (Safety Analysis Set) | Placebo (Safety Analysis Set)
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/88
Serious Adverse Events (participants affected / at risk) | 2/86 | 0/88
Other Adverse Events (participants affected / at risk) | 52/86 | 29/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTO-104 (Safety Analysis Set) (N=86) | Placebo (Safety Analysis Set) (N=88)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTO-104 (Safety Analysis Set) (N=86) | Placebo (Safety Analysis Set) (N=88)
Headache (Nervous system disorders) | 9 (86) | 7 (88)
Dizziness (Nervous system disorders) | 7 (7) | 4 (4)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (2)
Hypoesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Meniere's Disease (Ear and labyrinth disorders) | 5 (5) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 4 (4) | 2 (2)
Ear Pain (Ear and labyrinth disorders) | 3 (3) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Ear Discomfort (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Injection Site Pain (General disorders) | 2 (2) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT02717442/Prot_SAP_000.pdf